CLINICAL TRIAL: NCT06206083
Title: Molecular Classification in Mexican Patients With Endometrial Cancer and Its Impact on Prognosis
Status: Recruiting | Type: Observational
Sponsor: National Institute of Cancerología (Other Government)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, David Cantu, Doctor in Medical Sciences; Researcher in Medical Sciences, National Institute of Cancerología
Other Study IDs: (023/028/ICI/(CEI/017/23)
Record Dates: First submitted 2023-12-05; First posted 2024-01-16 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer; Prognostic factors
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Paraffin embeamed samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with EC endometroid: Patients with EC endometroid subtype and peripheral blood, treated during 2015-2019 at the INCan.
  Interventions: Genetic: Descriptive and analytical

INTERVENTIONS:
Genetic: Descriptive and analytical — Patients with EC endometroid

SUMMARY:
Endometrial cancer (EC) is one of the most common gynecological neoplasms, being the second in incidence and third in mortality in Mexico. Recent studies show that EC molecular classification (Cancer Genome Atlas Research Network, 2013) serves to establish a more accurate prognosis in these patients and regulate therapeutic behavior in a personalized manner. However, there are no studies on EC molecular classification in Mexican women or its impact on prognosis and the possible modification of targeted treatment. The investigators will determine the molecular classification in EC by next-generation sequencing (NGS) to detect TP53 and POLE somatic mutations, and immunohistochemical detection of microsatellite instability (MSH2, MLH1, PMS1, PMS2, MSH6, and MSH3) in a cohort of patients with endometrioid-type EC, endometrioid subtype, attended at the Instituto Nacional de Cancerología - Mexico (INCan) and determine its impact on clinical prognosis.

DETAILED DESCRIPTION:
The investigators will carry out a pilot study on patients with endometrioid type EC treated between 2015-2019. Samples of patients over 18 years of age admitted to the cohort with a diagnosis of endometrioid-type EC are already collected and will be evaluated for exome sequencing (N=32) and the detection of POLE mutations. DNA will be extracted using the "DNA/RNA AllPrep" kit (QIAGEN). Verification of adequate DNA extraction will be performed by quantifying using TapeStation (Agilent). Exome sequencing (N = 32 tumor samples and 32 somatic samples [leukocytes] from the same patient) will be carried out using Illumina's Nextera Rapid Capture Exome at Azenta Life Science (NJ, USA) following preset protocols and with a depth of 100X. The alignment and detection of variants will be done with the GATX-Mutect Suite (Broad Institute, USA) and the annotation of variant filtering with ANNOVAR. The identification of hotspots will be made according to Chen study. The immunohistochemistry (IHC) for microsatellite instability and overexpressed mutant TP53 (N = 94) will be done using established IHC protocols and will include MSH2, MLH1, PMS1, PMS2, MSH6, MSH3, and TP53.

ELIGIBILITY:
Criteria: Inclusion Criteria:

* Clinical diagnosis of endometrioid-type endometrial cancer with samples available
* That the patients have undergone surgery at INCan.

Exclusion Criteria:

* Samples with CEE of non-endometroid type.
* Samples from patients with double primary neoplasm, including carcinoma ductal in situ, squamous cell skin cancers, and cervical carcinoma in situ
* History of malignancy < 5 years prior with no evidence of disease (i.e., remission).

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — We will evaluate samples from females with endometrioid type EC t
Study Population: The investigators will evaluate samples from patients with endometrioid type EC treated between 2015-2019. Samples of patients over 18 years of age admitted to the cohort with a diagnosis of endometrioid-type EC are already collected and will be evaluated for exome sequencing (N=32) for the detection of POLE mutations.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
sequence the exome | 2024-2025
  Molecular classification of endometroid-type endometrial cancer in Mexican participants based on POLE and TP53 mutations as well as makers of microsatellite instability (MSH2, MLH1, PMS1, PMS2, MSH6, and MSH3).
Determine POLE mutations | 2024-2025
  Determine POLE mutations by massive next-generation sequencing of a discovery cohort in patients with endometroid-type EC.
Determine microsatellite instability | 2025-2026
  To perform validation of POLE mutation by real-time PCR in a validation cohort of patients with endometroid-type EC.
Validation | 2025-2026
  To perform validation of POLE mutation by real-time PCR in a validation cohort of patients with endometroid-type EC.

SECONDARY OUTCOMES:
Overall survival | 2025-2026
  To describe the overall survival of molecular types of endometroid-type EC in INCan patients.
Disease-free surviva | 2025-2026
  To describe the disease-free survival of the molecular types of endometroid-type EC in INCan patients.

CONTACTS AND LOCATIONS:
Overall Officials: David F Cantu-de-León, PhD, Principal Investigator — The Principal Investigator
Locations (1):
- Instituto Nacional de Cancerología, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Any time by direct request to the principal investigator
Access Criteria: Only for research purposes.